CLINICAL TRIAL: NCT02462473
Title: A Sequential and Parallel Cohort Design to Test the Clinical Utility of Antipsychotic Medication Levels in Plasma as Determined by Liquid Chromatography-Tandem Mass Spectrometry
Brief Title: A Study to Assess the Clinical Utility of Antipsychotic Medication Levels in Plasma as Determined by Liquid Chromatography-Tandem Mass Spectrometry
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor enrollment sponsor terminated early after enrolling 9 in Cohort 1 and no enrollment in Cohorts 2 and 3.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR106922; CODX0001NAP2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Aripiprazole; Olanzapine; Paliperidone; Quetiapine; Risperidone; Liquid Chromatography-Tandem Mass Spectrometry
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Aripiprazole; Olanzapine; Paliperidone Palmitate; Quetiapine Fumarate; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Participants will receive treatment as usual (TAU) which include one or more of the 5 antipsychotic medications (aripiprazole, olanzapine, paliperidone, quetiapine, and risperidone) for 12 weeks as determined by the treating clinician and the antipsychotic medication plasma level (AMPL) results will not be available to the clinicians until all participants in this cohort at a given site have completed their study participation.
  Interventions: Drug: Aripiprazole; Drug: Olanzapine; Drug: Paliperidone; Drug: Quetiapine; Drug: Risperidone
- Cohort 2 (Experimental): Participants will receive treatment as usual (TAU) which include one or more of the 5 antipsychotic medications (aripiprazole, olanzapine, paliperidone, quetiapine, and risperidone) for 12 weeks as determined by the treating clinician and the antipsychotic medication plasma level (AMPL) results will be provided to the clinician as they become available.
  Interventions: Drug: Aripiprazole; Drug: Olanzapine; Drug: Paliperidone; Drug: Quetiapine; Drug: Risperidone
- Cohort 3 (Experimental): Participants will receive treatment as usual (TAU) which include one or more of the 5 antipsychotic medications (aripiprazole, olanzapine, paliperidone, quetiapine, and risperidone) for 12 weeks as determined by the treating clinician and the antipsychotic medication plasma level (AMPL) results will not be available to the clinicians until all participants in cohorts 2 and 3 at a given site have completed participation in the active assessment phase.
  Interventions: Drug: Aripiprazole; Drug: Olanzapine; Drug: Paliperidone; Drug: Quetiapine; Drug: Risperidone

INTERVENTIONS:
Drug: Aripiprazole — Participants will receive aripiprazole at a dose of 5 milligram (mg) or higher, as oral formulation once daily for 12 weeks as part of participant treatment.
Drug: Olanzapine — Participants will receive olanzapine at a dose of 5 mg or higher, as oral formulation once daily for 12 weeks as part of participant treatment.
Drug: Paliperidone — Participants will receive paliperidone 3 mg or higher dose as oral formulation once daily or 39 mg or higher dose once every 4 weeks for 12 weeks as part of participant treatment.
Drug: Quetiapine — Participants will receive quetiapine at a dose of 150 mg or higher, as oral formulation once daily for 12 weeks as part of participant treatment.
Drug: Risperidone — Participants will receive risperidone 1 mg or higher dose, as oral formulation once daily or as injection of 12.5 mg or higher dose once every 2 weeks for 12 weeks as part of participant treatment.

SUMMARY:
The purpose of this study is to determine the number of Medication Treatment Modifications (MTMs) made by the clinician at every visit when antipsychotic medication plasma levels (AMPL) results are available compared to when AMPL results are not available.

DETAILED DESCRIPTION:
This is a naturalistic, open-label (all people know the identity of the intervention), multicenter (when more than one hospital or medical school team work on a medical research study), pilot clinical utility study with a sequential and parallel cohort design in participants with a diagnosis of schizophrenia or schizoaffective disorder. The study consists of up to 3 Phases: Screening Phase (Screening and first assessment visit should preferably take place on the same day), active assessment phase (12 weeks, An optional 12 week extension phase. Participants will be assigned to Cohort 1, or randomized to Cohort 2 or Cohort 3. Participants in cohorts 2 and 3 who are receiving long acting injectable (LAI) formulations of paliperidone and/or risperidone and complete participation in the active assessment phase) will have the option of continuing into the extension phase. The duration of study participation will be approximately 12 weeks. Participants in the optional extension phase will have an additional 12 weeks of study participation. The primary outcome will be measured by the number of Medication Treatment Modifications (MTMs) made by the clinician at every visit. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of schizophrenia (Code 295.90) or schizoaffective disorder (Code 295.70) according to Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM 5), based on history and clinical assessment by the investigator
* Participant has current active medication management issues and has experienced a medication treatment modification within the 6 weeks prior to Screening
* Participant is currently taking one or more of the following antipsychotic medications for at least 1 week for oral antipsychotics and at least 1 injection cycle for long-acting injectable (LAI) antipsychotics. In addition, the treating clinician plans to continue the antipsychotic medication(s) for at least 4 weeks subsequent to the Screening visit. Participant may be taking more than one formulation of a particular medication (such as oral and LAI) at or above the minimum dose specified in protocol. Qualifying formulations of the antipsychotic medications are: Aripiprazole (oral formulation only), Olanzapine (oral formulation only), Paliperidone (oral and/or LAI formulations), Quetiapine (oral formulation only), and Risperidone (oral and/or LAI formulations)
* Participant has had no clinically significant suicidal behavior or ideation during the week prior to Screening, according to the investigator's judgment
* Participant is generally healthy and has no clinically significant or unstable medical problems as determined by the investigator, except for the indication for which the antipsychotic treatment is being prescribed. This determination must be recorded in the participant's source documents and initialed by the investigator

Exclusion Criteria:

* Participant has been attending the outpatient psychiatric clinic for more than 12 months since the last psychiatric hospitalization
* During Screening, participant has active alcohol or substance use disorder (except tobacco) of moderate or severe severity according to DSM 5 criteria
* Participant has a history of or currently has a clinically significant (particularly unstable) medical illness, other than the indication for which the participant is taking antipsychotic therapy, that the investigator considers should exclude the participant or that could interfere with the participant completing the study or with interpretation of the study results. Treated, stable, chronic medical problems are allowed, as long as these conditions do not interfere with the study assessments
* Participant is receiving clozapine
* Participant has donated blood or blood products or had substantial loss of blood (ie, blood loss of approximately more than 450 milliliter (mL) or blood loss that required a blood transfusion) within 1 month of Screening or has the intention to donate blood or blood products during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (3):
- United States (3):
  - Torrance, California
  - Kissimmee, Florida
  - Conshohocken, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study had a planned enrollment of approximately 155 participants into 3 cohorts. However a total of 9 participants were enrolled and analyzed for efficacy and safety assessments in Cohort 1 and no participants were enrolled into Cohorts 2 or 3 of the study.
Groups:
- Cohort 1: Participants received treatment as usual (TAU) which include one or more of the 5 antipsychotic medications (aripiprazole, olanzapine, paliperidone, quetiapine, and risperidone) for 12 weeks.
Period: Overall Study
Arm/Group | Cohort 1
Started | 9
Completed | 5
Not Completed | 4
Not completed — Death | 1
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Arm/Group | Cohort 1
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (13.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Medication Treatment Modifications (MTM)
Description: Information on MTMs derived from data collected in the clinical assessment of the schizophrenia patient (CASP) questionnaire. The CASP captured changes in medications, changes in psychosocial treatments, visit frequency, and the need for any acute interventions. The CASP comprised of 3 sections covering several parameters. The CASP captured changes in treatment options which was used to compute MTM, as well as factors in clinical decision making and the influence of antipsychotic medication plasma levels (AMPL), when they were available, on clinical decision making.
Time Frame: Up to Week 12
Population: All enrolled participants who had a baseline CASP evaluation were included in the efficacy analysis set. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this endpoint.
Measure: Number; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 8
Participants | 4

2. Secondary Outcome: Clinical Global Impression-Severity (CGI-S) Score at Week 0 and 12
Description: Clinical Global Impression-Severity (CGI-S) rating scale used to rate the severity of a participant's overall clinical condition on a 7-point scale ranging from 1 (not ill) to 7 (extremely severe). Due to early study termination collected data was not summarized. Hence, individual data for each participant was reported.
Time Frame: Week 0, Week 12
Population: All enrolled participants who had a baseline CASP evaluation were included in the efficacy analysis set. One participant (Participant 4) was not analyzed at Week 12 due to discontinuation caused by death.
Measure: Number; unit: units on a scale
Arm/Group | Cohort 1
Number analyzed (Participants) | 9
units on a scale
  Participant 1 (Week 0) | 4
  Participant 1 (Week 12) | 3
  Participant 2 (Week 0) | 4
  Participant 2 (Week 12) | 3
  Participant 3 (Week 0) | 4
  Participant 3 (Week 12) | 4
  Participant 4 (Week 0) | 5
  Participant 5 (Week 0) | 3
  Participant 5 (Week 12) | 3
  Participant 6 (Week 0) | 3
  Participant 6 (Week 12) | 3
  Participant 7 (Week 0) | 3
  Participant 7 (Week 12) | 4
  Participant 8 (Week 0) | 4
  Participant 8 (Week 12) | 3
  Participant 9 (Week 0) | 3
  Participant 9 (Week 12) | 3

3. Secondary Outcome: Dimensions of Psychosis Symptom Severity Scale (DPSS) Total Score at Week 0 and 12
Description: The DPSS is a clinician-rated scale used to rate 8 domains commonly seen in patients with psychotic disorders. Each domain was rated on a 5-point scale (0 to 4) with anchored description of endpoints. Total score was computed by summing the scores of individual items (range of 0-32). Higher scores represent more severe condition. Due to early study termination collected data was not summarized. Hence, individual data for each participant was reported.
Time Frame: Week 0, Week 12
Population: as for outcome 2
Measure: Number; unit: units on a scale
Arm/Group | Cohort 1
Number analyzed (Participants) | 9
units on a scale
  Participant 1 (Week 0) | 12
  Participant 1 (Week 12) | 4
  Participant 2 (Week 0) | 8
  Participant 2 (Week 12) | 2
  Participant 3 (Week 0) | 8
  Participant 3 (Week 12) | 8
  Participant 4 (Week 0) | 14
  Participant 5 (Week 0) | 9
  Participant 5 (Week 12) | 4
  Participant 6 (Week 0) | 7
  Participant 6 (Week 12) | 4
  Participant 7 (Week 0) | 5
  Participant 7 (Week 12) | 8
  Participant 8 (Week 0) | 4
  Participant 8 (Week 12) | 4
  Participant 9 (Week 0) | 4
  Participant 9 (Week 12) | 6

4. Secondary Outcome: Antipsychotic Medication Plasma Levels (AMPL) During the Active Assessment Phase at Week 12
Description: AMPL of the individual participant during the active assessment phase was reported.
Time Frame: Week 12
Population: AMPL analysis set included all enrolled participants who had AMPL data for at least 1 visit. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this endpoint.
Measure: Number; unit: nanogram per milliliter
Arm/Group | Cohort 1
Number analyzed (Participants) | 8
nanogram per milliliter
  Participant 1- ARIPIPRAZOLE | 596.00
  Participant 1- DEHYDROARIPIPRAZOLE | 139.00
  Participant 2- OLANZAPINE | 27.30
  Participant 2- PALIPERIDONE | 45.10
  Participant 3- 7-OH QUETIAPINE | 43.10
  Participant 3-NORQUETIAPINE | 660.00
  Participant 3-QUETIAPINE | 280.00
  Participant 3-QUETIAPINE SULFOXIDE | 660.00
  Participant 5-7-OH QUETIAPINE | 7.72
  Participant 5-NORQUETIAPINE | 153.00
  Participant 5-QUETIAPINE | 50.30
  Participant 5-QUETIAPINE SULFOXIDE | 321.00
  Participant 6-ARIPIPRAZOLE | 464.00
  Participant 6-DEHYDROARIPIPRAZOLE | 112.00
  Participant 7-PALIPERIDONE | 31.00
  Participant 7-RISPERIDONE | 26.20
  Participant 8-ARIPIPRAZOLE | 168.00
  Participant 8-DEHYDROARIPIPRAZOLE | 33.00
  Participant 9- 7-OH QUETIAPINE | 0.200
  Participant 9- NORQUETIAPINE | 2.00
  Participant 9- PALIPERIDONE | 0.100
  Participant 9- QUETIAPINE | 2.00
  Participant 9- QUETIAPINE SULFOXIDE | 2.00
  Participant 9- RISPERIDONE | 0.100

5. Secondary Outcome: Number of Participants With Factors Considered in Clinical Decision as Assessed by Clinical Assessment of the Schizophrenia Patient (CASP)
Description: The CASP and data on concomitant medications and psychosocial treatments were used to evaluate the impact of AMPL results on other aspects of clinical decision making.
Time Frame: Up to Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 6
participants
  Side Effects Of Medication | 3
  Attitude Toward Treatment | 2
  Report of Increased Symptoms | 4
  Report of Decrease in Symptoms | 3
  Patient Still Symptomatic | 1
  Patient Ideation | 1

6. Secondary Outcome: Clinician's Rating Scale of Adherence (CRS) Score at Week 0 and 12
Description: The CRS is an ordinal scale filled by the clinician. The scores range from 1 to 7 that were used to quantify the clinician's assessment of treatment adherence by the patient. Higher scores indicate greater adherence. Due to early study termination collected data was not summarized. Hence, individual data for each participant was reported.
Time Frame: Week 0, Week 12
Population: as for outcome 2
Measure: Number; unit: units on a scale
Arm/Group | Cohort 1
Number analyzed (Participants) | 9
units on a scale
  Participant 1 (Week 0) | 7
  Participant 1 (Week 12) | 7
  Participant 2 (Week 0) | 7
  Participant 2 (Week 12) | 7
  Participant 3 (Week 0) | 7
  Participant 3 (Week 12) | 7
  Participant 4 (Week 0) | 7
  Participant 5 (Week 0) | 7
  Participant 5 (Week 12) | 7
  Participant 6 (Week 0) | 7
  Participant 6 (Week 12) | 7
  Participant 7 (Week 0) | 7
  Participant 7 (Week 12) | 7
  Participant 8 (Week 0) | 7
  Participant 8 (Week 12) | 7
  Participant 9 (Week 0) | 7
  Participant 9 (Week 12) | 7

7. Secondary Outcome: Adherence to Antipsychotic Medication as Assessed by Brief Adherence Rating Scale (BARS) at Week 0 and 12
Description: The BARS is a 4-item scale that includes 3 questions and an overall visual analog rating scale that assesses participant's knowledge about his/her medication. The key measure of adherence is the visual analog scale and assesses the percentage of doses taken by the participants in the past month (0 percent [%] - 100%). The 3 questions include: number of prescribed doses per day, number of days in the past month when the participant did not take the prescribed doses, and the number of days in the past month when the participant took less than the prescribed dose. Due to early study termination collected data was not summarized. Hence, individual data for each participant was reported.
Time Frame: Week 0, Week 12
Population: as for outcome 2
Measure: Number; unit: percent adherence
Arm/Group | Cohort 1
Number analyzed (Participants) | 9
percent adherence
  Participant 1 (Week 0) | 100
  Participant 1 (Week 12) | 100
  Participant 2 (Week 0) | 100
  Participant 2 (Week 12) | 100
  Participant 3 (Week 0) | 100
  Participant 3 (Week 12) | 100
  Participant 4 (Week 0) | 97
  Participant 5 (Week 0) | 93
  Participant 5 (Week 12) | 90
  Participant 6 (Week 0) | 90
  Participant 6 (Week 12) | 96
  Participant 7 (Week 0) | 90
  Participant 7 (Week 12) | 95
  Participant 8 (Week 0) | 100
  Participant 8 (Week 12) | 100
  Participant 9 (Week 0) | 100
  Participant 9 (Week 12) | 100

8. Secondary Outcome: Patient Satisfaction Survey (PSS) Total Score at Week 0 and 12
Description: The PSS is a brief scale designed to capture a psychiatric patient's satisfaction with a clinician. The scale covers 6 domains: Trust (3 items), Communication (3 items), Exploration of Ideas/Options (2 items), Body Language (2 items), Active Listening (4 items), and Miscellaneous Items (6 items). Out of the 20 items, the first 19 are scored on a 5-point Likert Scale (1=strongly disagree, 2=disagree, 3=satisfactory, 4=agree, 5=strongly agree). The last question (6f) is a free-response question asking for input on how the clinician might improve. Sum of scores of individual items give a total score (range 9-95). Higher scores indicate greater degree of satisfaction. Due to early study termination collected data was not summarized. Hence, individual data for each participant was reported.
Time Frame: Week 0, Week 12
Population: as for outcome 2
Measure: Number; unit: units on a scale
Arm/Group | Cohort 1
Number analyzed (Participants) | 9
units on a scale
  Participant 1 (Week 0) | 76
  Participant 1 (Week 12) | 76
  Participant 2 (Week 0) | 52
  Participant 2 (Week 12) | 57
  Participant 3 (Week 0) | 57
  Participant 3 (Week 12) | 57
  Participant 4 (Week 0) | 48
  Participant 5 (Week 0) | 66
  Participant 5 (Week 12) | 64
  Participant 6 (Week 0) | 76
  Participant 6 (Week 12) | 76
  Participant 7 (Week 0) | 76
  Participant 7 (Week 12) | 72
  Participant 8 (Week 0) | 63
  Participant 8 (Week 12) | 72
  Participant 9 (Week 0) | 71
  Participant 9 (Week 12) | 76

ADVERSE EVENTS:
Arm/Group | Cohort 1
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=9)
Death (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=9)
External ear inflammation (Ear and labyrinth disorders) | 1
Pharyngitis (Infections and infestations) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Miliaria (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Due to poor enrollment, the study was terminated early by the sponsor after enrolling only 9 participants in Cohort 1 and no participants were enrolled in Cohorts 2 and 3.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.